CLINICAL TRIAL: NCT05140382
Title: A Modular Phase II, Open-label, Multicentre Study to Assess AZD4573 Efficacy and Safety as Monotherapy or in Combination With Anti-cancer Agents in Patients With Relapsed/Refractory Peripheral T-cell Lymphoma or Classical Hodgkin Lymphoma
Brief Title: AZD4573 as Monotherapy or in Combinations With Anti-cancer Agents in Patients With r/r PTCL or r/r cHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8231C00001; 2021-002570-54 (EudraCT Number)
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-07

CONDITIONS: Relapsed/Refractory Peripheral T-cell Lymphoma; Relapsed/Refractory Classical Hodgkins Lymphoma
Keywords: AZD4573; Modular study; Dose confirmation; Dose expansion
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD4573 (Monotherapy) (Experimental): Eligible participants with either r/r PTCL, r/r NKTCL or r/r cHL will receive AZD4573 as monotherapy.
  Interventions: Drug: AZD4573

INTERVENTIONS:
Drug: AZD4573 — AZD4573 will be given intravenously

SUMMARY:
This is a modular dose confirmation and expansion study. The core study design is to assess the efficacy of AZD4573, administered as monotherapy or combination therapy, to participants with either r/r PTCL or r/r cHL and to confirm the safety profiles and PK in these populations. Module 1 of this study will evaluate the efficacy, safety, and tolerability of AZD4573 monotherapy in participants with r/r PTCL or r/r cHL. If AZD4573 monotherapy is found to have promising anti-tumour efficacy in Module 1, an AZD4573 monotherapy Phase II expansion may be added via a substantial protocol amendment.

DETAILED DESCRIPTION:
Module 1 will consist of two r/r PTCL cohorts and one cHL cohort; and each cohort includes 21 participants. A comprehensive initial review of all safety and PK/PD data will be conducted in approximately the first 6 participants of each cohort (safety run-in), with separate Safety Review Committees (SRCs) for each cohort executed independently. The safety assessment will be undertaken by the SRC. Each cohort will have a separate dose confirmation, assessed independently by the SRC, to assess safety and PK/PD data compared to the known profiles in the first time in human study (Study D8230C00001) lymphoma population. These SRC reviews will confirm whether the recommended phase II dose for lymphoma (IV infusion 12 mg once weekly, including intra-participant ramp-up) is safe and tolerable or if additional dose optimisation is indicated at a revised dose and/or schedule. All cohorts can be opened and delivered independently of each other.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed with one of the following, as defined by the World Health Organisation:

  * Peripheral T-cell Lymphoma
  * Classical Hodgkin Lymphoma
* Eastern Cooperative Oncology Group performance status of ≤ 2.
* Must have received at least 1 prior line of therapy for the treatment of current disease and have documented relapsed or refractory active disease requiring treatment, defined as:

  * Recurrence of disease after response to prior line(s) of therapy, or
  * Progressive disease after completion of or on the treatment regimen preceding entry into the study, or
  * Disease which did not achieve an objective response (CR or PR).
* Uric acid level < ULN at screening. If hyperuricaemia is present at screening, SoC therapy should be administered (including IV fluid and rasburicase or allopurinol) to reduce the uric acid levels to < ULN before the start of study intervention.
* Willing and able to participate in all required evaluations and procedures in this study protocol including receiving IV administration of study drug and being admitted, if required, for at least 24 hours during study drug administration.
* Fresh tumour tissue or archival tumour tissue must be confirmed to be available at screening.
* Adequate haematologic function at screening.
* PTCL Only: All participants with PTCL must be willing and able to provide baseline bone marrow aspirate and/or biopsy no older than 3 months and agree to undergo post-treatment bone marrow biopsy when required to confirm response.

Additional Module 1 Inclusion Criteria

Prior lines of therapy:

* PTCL: Participants must have failed at least 1 prior therapy for the treatment of PTCL.

  * Non NK-PTCL (Cohort 1): Prior therapy must have included an alkylating agent and/or anthracycline. In addition, ALCL participants must have received brentuximab vedotin (BV) as part of prior therapy.
  * NKTCL (Cohort 2): Prior treatment must have included a platinum agent and/or asparaginase.
* cHL (Cohort 3): Participants must have failed at least 2 prior therapies for the treatment of cHL (including BV and anti-PD1) except where unable to receive BV or anti-PD1 due to neuropathy or autoimmune disease.
* Presence of at least 1 radiographically measurable, FDG-avid lymphoma disease lesion > 1.5 cm (according to the Lugano (2014) criteria [Cheson et al 2014]).

Exclusion Criteria

Type of Participant and Disease Characteristics:

* PTCL only: Presence of bulky disease (defined as largest lymphoma lesion ≥ 10 cm) or a LDH value > 3 x ULN.
* PTCL only: Diagnosis of any of the following: Lymphoblastic/precursor T-cell lymphoma or leukaemia; T-cell prolymphocytic leukaemia; T-cell large granular lymphocytic leukaemia; Cutaneous T-cell lymphoma (eg, primary cutaneous type ALCL, mycosis fungoide/Sezary syndrome).

Medical Conditions:

* With the exception of alopecia and neuropathy, presence of any unresolved non haematological toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment.
* Presence of, or history of, CNS lymphoma, leptomeningeal disease, or spinal cord compression.
* History of prior non-haematological malignancy except for the following:

  * Malignancy treated with curative intent and with no evidence of active disease present for more than 1 year prior to screening and felt to be at low risk for recurrence by treating physician.
  * Adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled non-melanomatous skin cancer.
  * Adequately treated carcinoma in situ without current evidence of disease.
* Any evidence of:

  * Severe or uncontrolled systemic disease (eg, severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease]).
  * Current unstable or uncompensated respiratory or cardiac conditions.
  * Uncontrolled hypertension.
  * Uncontrolled active systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
  * IV anti-infective treatment within 1 week before first dose of study drug.
* Known history of infection with HIV.
* Serologic status reflecting active hepatitis B or C infection:

  * Participants who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative PCR result before enrolment. Those who are hepatitis B surface antigen positive or hepatitis B PCR-positive will be excluded.
  * Participants who are hepatitis C antibody positive will need to have a negative PCR result before enrolment. Those who are hepatitis C PCR-positive will be excluded.
* Any of the following cardiac criteria:

  * Resting QT interval corrected using Fridericia's formula (QTcF) ≥ 470 msec obtained from a single ECG.
  * Any clinically important abnormalities in rhythm (except for participants with a pacemaker in place), conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block).
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age.
* Documented confirmation and ongoing treatment of adrenal gland insufficiency or pancreatitis.
* Undergone any of the following procedures or experienced any of the following conditions within 6 months prior to first dose:

  * Coronary artery bypass graft
  * Angioplasty
  * Vascular stent
  * Myocardial infarction
  * Angina pectoris
  * CHF (New York Heart Association Class ≥ 2)
  * Ventricular arrhythmias requiring continuous therapy
  * Atrial fibrillation, which is judged as uncontrolled by the treating physician
  * Haemorrhagic or thrombotic stroke, including transient ischemic attacks or any other CNS bleeding

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (6):
  - Research Site, Duarte, California
  - Research Site, Boston, Massachusetts
  - Research Site, Hackensack, New Jersey
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
- Australia (3):
  - Research Site, Clayton
  - Research Site, Melbourne
  - Research Site, Nedlands
- France (5):
  - Research Site, Besançon
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, Lille
  - Research Site, Montpellier
- Italy (2):
  - Research Site, Bologna
  - Research Site, Napoli
- Research Site, Seoul, South Korea
- Research Site, Lund, Sweden
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (2):
  - Research Site, Headington
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8231C00001&attachmentIdentifier=2741dd3d-4ffa-4449-b693-3f33ed4fa400&fileName=Protocol_Amendment_Main_2.0_English__D8231C00001_final_Redacted_Sponsor_approved_pdfa.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8231C00001&attachmentIdentifier=3b65d7e9-bb44-413d-bae5-c8611c498bd5&fileName=Statistical_Analysis_Plan_12_Dec_2023_D8231C00001_final_Redacted_Sponsor_approved_pdfa.pdf&versionIdentifier=
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8231C00001&attachmentIdentifier=67fd798e-7117-43c4-a149-e0bb2bfa67be&fileName=CSR_Synopsis_D8231C00001_Draft_2_to_sponsor_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 15 December 2021 and completed on 16 February 2024. The study was conducted at 27 sites in 7 countries worldwide (Australia, France, Italy, South Korea, Taiwan, United Kingdom and United States).
Pre-assignment Details: Participants who met the inclusion criteria and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
Groups:
- Cohort 1 Non-natural Killer Peripheral T-cell Lymphoma (Non NK PTCL): Participants with non-NK PTCL received 12 mg dose of AZD4573 once weekly until disease progression.
- Cohort 2 Natural Killer T-cell Lymphoma (NK PTCL): Participants with NK PTCL received 12 mg dose of AZD4573 once weekly until disease progression.
- Cohort 3 Classical Hodgkins Lymphoma (cHL): Participants with cHL received 12 mg dose of AZD4573 once weekly until disease progression.
Period: Overall Study
Arm/Group | Cohort 1 Non-natural Killer Peripheral T-cell Lymphoma (Non NK PTCL) | Cohort 2 Natural Killer T-cell Lymphoma (NK PTCL) | Cohort 3 Classical Hodgkins Lymphoma (cHL)
Started | 31 | 2 | 19
Completed | 0 | 0 | 0
Not Completed | 31 | 2 | 19
Not completed — Death | 3 | 0 | 0
Not completed — Investigator decision | 1 | 0 | 0
Not completed — Other | 4 | 0 | 1
Not completed — Progressive disease | 20 | 1 | 12
Not completed — Subjective disease progression | 2 | 1 | 0
Not completed — Unknown at data cut-off | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 4
Not completed — Withdrawal of consent | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included for baseline characteristics and it included all participants who received any amount of any study intervention.
Groups:
- Cohort 1 Non-NK PTCL: Participants with non-NK PTCL received 12 mg dose of AZD4573 once weekly until disease progression.
- Cohort 2 NK PTCL: Participants with NK PTCL received 12 mg dose of AZD4573 once weekly until disease progression.
- Cohort 3 cHL: Participants with cHL received 12 mg dose of AZD4573 once weekly until disease progression.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL | Total
Number analyzed (Participants) | 31 | 2 | 19 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (12.2) | 61.0 (8.5) | 46.5 (14.7) | 55.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 0 | 10 | 23
  Male | 18 | 2 | 9 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 2 | 0 | 2 | 4
  Race: Asian | 3 | 2 | 6 | 11
  Race: White | 18 | 0 | 7 | 25
  Race: Other | 1 | 0 | 1 | 2
  Race: Not reported | 2 | 0 | 2 | 4
  Race: Missing | 5 | 0 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 4 | 0 | 0 | 4
  Ethnicity: Not Hispanic or Latino | 20 | 2 | 16 | 38
  Ethnicity: Missing | 7 | 0 | 2 | 9
  Ethnicity: Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the proportion of participants who have a tumour response of complete response [CR] or partial response [PR] according to the Lugano (2014) response criteria for malignant lymphoma.
Time Frame: From Screening (Day -30 to Day-1) until disease progression or survival until death (26 months)
Population: Response evaluable set included all dosed participants who had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 31 | 2 | 19
Percentage of participants | 22.6 [9.59 to 41.10] | 0 [0 to 84.19] | 21.1 [6.05 to 45.57]

2. Secondary Outcome: Complete Response (CR) Rate
Description: Complete response rate is defined as proportion of participants who have a complete response according to the Lugano (2014) response criteria.
Time Frame: From Screening (Day -30 to Day-1) until disease progression or survival until death (26 months).
Population: Response evaluable set included all dosed participants who had measurable disease at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 31 | 2 | 19
Percentage of participants | 19.4 | 0 | 15.8

3. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response is defined as the time from the first objective response to the time of documented disease progression or death due to any cause, whichever occurs first.
Time Frame: From Screening (Day -30 to Day-1) until disease progression or survival until death (26 months).
Population: Response evaluable set included all dosed participants who have measurable disease at baseline and had objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 7 | 0 | 4
Months | NA [1.8 to NA] — The median and 95% CI were calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and were non estimable as there was insufficient number of participants with the event of interest (less than 50%) occurred in the study. |  | 5.2 [1.9 to NA] — The 95% CI was calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and was non estimable as there was insufficient number of participants with the event of interest (less than 50%) occurred in the study.

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from the date of first dose to documented disease progression, or death from any cause, whichever occurs first.
Time Frame: From Screening (Day -30 to Day-1) until disease progression or survival until death (26 months).
Population: Full analysis set included all participants who received any amount of any study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 31 | 2 | 19
Months | 1.8 [1.51 to 2.17] | 0.7 [0.66 to NA] — Here, "NA" indicates that higher limit of 95% CI could not be evaluated due to smaller number of participants. | 1.9 [1.64 to 4.11]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of first dose to death from any cause.
Time Frame: From Screening (Day -30 to Day-1) until disease progression or survival until death (26 months).
Population: Full analysis set included all participants who received any amount of any study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 31 | 2 | 19
Months | 8.6 [2.33 to 10.18] | NA [0.66 to NA] — Here, "NA" indicates that median and higher limit of 95% CI could not be evaluated due to smaller number of participants. | NA [10.05 to NA] — Here "NA" indicates that the median and upper limit of 95% CI could not be calculated due to less number of events of interest (less than 50%).

6. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious AEs (SAE)
Description: The safety and tolerability of AZD4573 was assessed.
Time Frame: From treatment period (Cycle 1) to follow up visit (30 [± 7] ) days from the last dose (upto 26 months).
Population: Safety set included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 31 | 2 | 19
Participants
  Any AE | 31 | 2 | 18
  Any AE possibly related to treatment | 31 | 2 | 16
  Any AE of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher | 29 | 2 | 15
  Any AE of CTCAE grade 3 or higher, possibly related to treatment | 27 | 2 | 13
  Any AE with outcome = death | 2 | 1 | 0
  Any AE with outcome = death, possibly related to treatment | 2 | 0 | 0
  Any SAE (including events with outcome = death) | 21 | 2 | 11
  Any SAE (including events with outcome = death), possibly related to treatment | 16 | 1 | 8

7. Secondary Outcome: Maximum Observed Plasma (Peak) Drug Concentration (Cmax)
Description: The plasma PK of AZD4573 when administered in participants was assessed.
Time Frame: Cycle 1 (Cycle length is 35 days), Day 1 of Weeks 1-3 and Cycle 2 (Cycle length is 21 Days), Day 1.
Population: Pharmacokinetic (PK) set included all participants who received any amount of study intervention with at least 1 reportable concentration. Here, 'n" (number analyzed in each row) signifies the participants with available data that were analyzed for each timepoint of this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 31 | 2 | 19
Nanogram per milliliter (ng/mL)
  Cycle 1 week 1 day 1 | 159.9 (53.2) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 201.8 (82.1)
  Cycle 1 week 2 day 1: number analyzed (Participants) | 25 | 1 | 15
  Cycle 1 week 2 day 1 | 312.4 (84.5) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 278.2 (73.8)
  Cycle 1 week 3 day 1: number analyzed (Participants) | 25 | 1 | 16
  Cycle 1 week 3 day 1 | 265.5 (54.1) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 376.3 (89.9)
  Cycle 2 day 1: number analyzed (Participants) | 16 | 0 | 14
  Cycle 2 day 1 | 308.6 (65.9) |  | 381.8 (82.5)

8. Secondary Outcome: Area Under the Plasma Concentration Curve From Zero to the Last Quantifiable Concentration (AUClast)
Description: The plasma PK of AZD4573 when administered in participants was assessed.
Time Frame: Cycle 1 (Cycle length is 35 days), Day 1 of Weeks 1-3 and Cycle 2 (Cycle length is 21 Days), Day 1.
Population: PK set included all participants who received any amount of study intervention with at least 1 reportable concentration. Here, 'n" (number analyzed in each row) signifies the participants with available data that were analyzed for each timepoint of this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)*ng/mL
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 31 | 2 | 19
hours (h)*ng/mL
  Cycle 1 week 1 day 1 | 913.3 (95.0) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 1039 (113.5)
  Cycle 1 week 2 day 1: number analyzed (Participants) | 25 | 1 | 15
  Cycle 1 week 2 day 1 | 1695 (102.3) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 1646 (86.7)
  Cycle 1 week 3 day 1: number analyzed (Participants) | 25 | 1 | 16
  Cycle 1 week 3 day 1 | 1651 (76.5) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 2228 (75.0)
  Cycle 2 day 1: number analyzed (Participants) | 16 | 0 | 14
  Cycle 2 day 1 | 1933 (81.2) |  | 2083 (115.9)

9. Secondary Outcome: Area Under Plasma Concentration Time Curve From Zero to Infinity (AUC0-inf) of AZD4573
Description: The plasma PK of AZD4573 when administered in participants was assessed.
Time Frame: Cycle 1 (Cycle length is 35 days), Day 1 of Weeks 1-3 and Cycle 2 (Cycle length is 21 Days), Day 1.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 18 | 1 | 12
h*ng/mL
  Cycle 1 week 1 day 1: number analyzed (Participants) | 18 | 0 | 9
  Cycle 1 week 1 day 1 | 1294 (82.9) |  | 1872 (59.3)
  Cycle 1 week 2 day 1: number analyzed (Participants) | 17 | 1 | 9
  Cycle 1 week 2 day 1 | 1711 (86.8) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 1984 (62.9)
  Cycle 1 week 3 day 1 | 1490 (71.5) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 2643 (88.2)
  Cycle 2 day 1: number analyzed (Participants) | 14 | 0 | 7
  Cycle 2 day 1 | 1885 (72.9) |  | 1899 (89.0)

10. Secondary Outcome: Time to Reach Peak Observed Concentration Following Drug Administration (Tmax)
Description: The plasma PK of AZD4573 when administered in participants was assessed.
Time Frame: Cycle 1 (Cycle length is 35 days), Day 1 of Weeks 1-3 and Cycle 2 (Cycle length is 21 Days), Day 1.
Population: as for outcome 8
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 31 | 2 | 19
Hour
  Cycle 1 week 1 day 1 | 2.000 [0.97 to 6.00] | NA [1.90 to 2.15] — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 2.083 [1.00 to 23.00]
  Cycle 1 week 2 day 1: number analyzed (Participants) | 25 | 1 | 15
  Cycle 1 week 2 day 1 | 2.083 [1.87 to 6.08] | NA [2.15 to 2.15] — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 2.083 [1.87 to 6.00]
  Cycle 1 week 3 day 1: number analyzed (Participants) | 25 | 1 | 16
  Cycle 1 week 3 day 1 | 2.083 [0.87 to 6.00] | NA [2.25 to 2.25] — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 2.133 [1.78 to 4.00]
  Cycle 2 day 1: number analyzed (Participants) | 16 | 0 | 14
  Cycle 2 day 1 | 2.133 [1.00 to 3.58] |  | 2.083 [0.97 to 5.02]

11. Secondary Outcome: Half-life (t1/2) of AZD4573
Description: The plasma PK of AZD4573 when administered in participants was assessed.
Time Frame: Cycle 1 (Cycle length is 35 days), Day 1 of Weeks 1-3 and Cycle 2 (Cycle length is 21 Days), Day 1.
Population: as for outcome 8
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 18 | 1 | 12
Hour
  Cycle 1 week 1 day 1: number analyzed (Participants) | 18 | 0 | 9
  Cycle 1 week 1 day 1 | 5.772 [1.67 to 11.6] |  | 5.858 [3.68 to 7.90]
  Cycle 1 week 2 day 1: number analyzed (Participants) | 17 | 1 | 9
  Cycle 1 week 2 day 1 | 5.448 [4.10 to 11.3] | NA [6.80 to 6.80] — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 5.250 [4.11 to 9.71]
  Cycle 1 week 3 day 1 | 5.435 [1.15 to 10.5] | NA [5.09 to 5.09] — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 5.499 [3.93 to 23.5]
  Cycle 2 day 1: number analyzed (Participants) | 14 | 0 | 7
  Cycle 2 day 1 | 6.669 [3.50 to 16.0] |  | 4.323 [3.56 to 14.7]

12. Secondary Outcome: Systematic Clearance (CL)
Description: The plasma PK of AZD4573 when administered in participants was assessed.
Time Frame: Cycle 1 (Cycle length is 35 days), Day 1 of Weeks 1-3 and Cycle 2 (Cycle length is 21 Days), Day 1.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 18 | 1 | 11
Liter/hour
  Cycle 1 week 1 day 1: number analyzed (Participants) | 18 | 0 | 9
  Cycle 1 week 1 day 1 | 4.636 (82.9) |  | 3.205 (59.3)
  Cycle 1 week 2 day 1: number analyzed (Participants) | 17 | 1 | 9
  Cycle 1 week 2 day 1 | 5.137 (82.3) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 4.537 (62.9)
  Cycle 1 week 3 day 1 | 7.799 (69.5) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 4.965 (74.7)
  Cycle 2 day 1: number analyzed (Participants) | 14 | 0 | 7
  Cycle 2 day 1 | 6.367 (72.9) |  | 6.064 (85.9)

13. Secondary Outcome: Volume of Distribution at Terminal Phase (Vz)
Description: The plasma PK of AZD4573 when administered in participants was assessed.
Time Frame: Cycle 1 (Cycle length is 35 days), Day 1 of Weeks 1-3 and Cycle 2 (Cycle length is 21 Days), Day 1.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 18 | 1 | 11
Liter
  Cycle 1 week 1 day 1: number analyzed (Participants) | 18 | 0 | 9
  Cycle 1 week 1 day 1 | 38.59 (49.0) |  | 26.45 (54.2)
  Cycle 1 week 2 day 1: number analyzed (Participants) | 17 | 1 | 9
  Cycle 1 week 2 day 1 | 45.96 (53.8) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 37.68 (37.5)
  Cycle 1 week 3 day 1 | 58.92 (33.1) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 44.34 (55.7)
  Cycle 2 day 1: number analyzed (Participants) | 14 | 0 | 7
  Cycle 2 day 1 | 63.45 (41.6) |  | 43.38 (59.0)

14. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: The plasma PK of AZD4573 when administered in participants was assessed.
Time Frame: Cycle 1 (Cycle length is 35 days), Day 1 of Weeks 1-3 and Cycle 2 (Cycle length is 21 Days), Day 1.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
Number analyzed (Participants) | 18 | 1 | 11
Liter
  Cycle 1 week 1 day 1: number analyzed (Participants) | 18 | 0 | 9
  Cycle 1 week 1 day 1 | 35.80 (51.1) |  | 24.20 (54.3)
  Cycle 1 week 2 day 1: number analyzed (Participants) | 17 | 1 | 9
  Cycle 1 week 2 day 1 | 39.25 (51.3) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 33.20 (36.9)
  Cycle 1 week 3 day 1 | 50.32 (27.8) | NA (NA) — Here, "NA" indicates that data could not be evaluated due to smaller number of participants. | 37.99 (66.3)
  Cycle 2 day 1: number analyzed (Participants) | 14 | 0 | 7
  Cycle 2 day 1 | 55.93 (36.8) |  | 37.29 (54.6)

ADVERSE EVENTS:
Time Frame: From treatment period (Cycle 1) to follow up visit (30 [± 7] ) days from the last dose (upto 26 months).
Arm/Group | Cohort 1 Non-NK PTCL | Cohort 2 NK PTCL | Cohort 3 cHL
All-Cause Mortality (participants affected / at risk) | 17/31 | 1/2 | 2/19
Serious Adverse Events (participants affected / at risk) | 21/31 | 2/2 | 11/19
Other Adverse Events (participants affected / at risk) | 31/31 | 2/2 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Non-NK PTCL (N=31) | Cohort 2 NK PTCL (N=2) | Cohort 3 cHL (N=19)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Fanconi syndrome acquired (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 2 (9) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Non-NK PTCL (N=31) | Cohort 2 NK PTCL (N=2) | Cohort 3 cHL (N=19)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 11 (21) | 0 (0) | 10 (15)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 1 (7)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 24 (126) | 1 (1) | 13 (54)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (43) | 1 (1) | 4 (9)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (2) | 0 (0)
Serum sickness (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 2 (5)
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 (9) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (16) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (14) | 1 (1) | 4 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (8) | 0 (0) | 2 (3)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (4) | 0 (0) | 4 (6)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 12 (18) | 0 (0) | 7 (8)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (14) | 1 (1) | 9 (14)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 8 (10) | 0 (0) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 1 (1)
Skin weeping (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site thrombosis (General disorders) | 3 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 6 (6)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (3) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (16) | 1 (1) | 3 (5)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 19 (90) | 1 (1) | 11 (35)
Amylase increased (Investigations) | 3 (6) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 21 (101) | 2 (3) | 11 (42)
Bilirubin conjugated increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 3 (5) | 0 (0) | 2 (5)
Blood bilirubin increased (Investigations) | 14 (46) | 2 (2) | 5 (18)
Blood calcium decreased (Investigations) | 1 (4) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (3) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood fibrinogen increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 3 (4) | 0 (0) | 0 (0)
Blood phosphorus increased (Investigations) | 4 (6) | 0 (0) | 2 (5)
Blood potassium decreased (Investigations) | 2 (5) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 3 (4) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 10 (18) | 0 (0) | 4 (7)
International normalised ratio increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (4) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 2 (2) | 0 (0) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Troponin increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 6 (34) | 0 (0) | 1 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT05140382/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT05140382/SAP_001.pdf